CLINICAL TRIAL: NCT01733433
Title: Influence of Taping on Postural Control in Subjects With Chronic Ankle Instability (CAI).
Brief Title: Influence of Taping on Postural Control in Subjects With Chronic Ankle Instability
Acronym: CAI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2012/480
Record Dates: First submitted 2012-11-13; First posted 2012-11-27 (Estimated); Last update posted 2021-12-02 (Actual); Status verified 2021-11

CONDITIONS: Chronic Ankle Instability

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- taped ankle (Experimental): Subjects will be taped in at the ankle for a series of exercises.
  Interventions: Procedure: Taping the ankle

INTERVENTIONS:
Procedure: Taping the ankle — Subjects will be taped in at the ankle for performing several exercises.

SUMMARY:
The main goal of this study is to evaluate the effect of taping on postural control during dynamic exercises. 30 subjects with Chronic ankle instability (CAI) will be included in the study. Several questionnaires regarding anthropometric data, medical history, activity level and functional status will be filled in by the participants. Postural control will be measured using a force plate and an optoelectronic system to capture lower limb kinematics. Subjects will be asked to perform a forward hop, sideward hop and a vertical drop, and they have to maintain their balance for 10 seconds after landing. 5 good trials of each movement will be captured. Subjects with CAI will perform these exercises with and without tape. Hypothesis is that subjects with CAI that tape will enhance postural control.

ELIGIBILITY:
Inclusion Criteria:

* a history of at least one ankle sprain which resulted in pain, swelling and stiffness, prohibiting participation in sport-, recreational or other activities for at least 3 weeks
* repeated ankle sprains
* presence of giving way
* feeling of weakness around the ankle
* a decreased functional participation (recreational, competitive or professionally)

Exclusion Criteria:

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2015-02 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Immediate postural control with tape on ankle. | for 75 minutes, the duration of the exercises.
  Postural control will be measured using a force plate and an optoelectronic system to capture lower limb kinematics.

SECONDARY OUTCOMES:
Subjective evaluation of the effect of taping on pain | 1 minute after the exercises (which last approximately 75 minutes).
  Evaluation will be done using a VAS scale.
Subjective evaluation of the effect of taping on difficulty level. | 1 minute after the exercises (which last approximately 75 minutes).
  This will be evaluated by interviewing the subject.
Subject evaluation of the effect of taping on instability feelings. | 1 minute after the exercises (which last approximately 75 minutes).
  This will be evaluated by interviewing the subject.

CONTACTS AND LOCATIONS:
Overall Officials: Philip Roosen, PhD, Principal Investigator — University Ghent
Locations (1):
- Ghent University, Ghent, Belgium